CLINICAL TRIAL: NCT04648735
Title: Driving Evaluation and Fitness for Persons With Cognitive Impairments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Ling-Hui Chang, Associate Professor, National Cheng Kung University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: National ChengKung University
Record Dates: First submitted 2020-11-22; First posted 2020-12-01 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Mild Cognitive Impairment; Dementia, Mild; Driving Impaired; Drive
Keywords: Mild Cognitive Impairment; dementia; driving fitness; driving rehabilitation
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: an observational, cross-sectional research design
Who Masked: Participant, Outcomes Assessor
Masking Description: the participant and the outcome assessor were both blind to the design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drivers with cognitive impairments (Experimental): The participants firstly completed a questionnaire of driving history and perceived driving competence, followed with a clinical physical and cognitive-perceptual assessment battery conducted by an occupational therapist to note any potential deficits that might affect driving performance. The participants, on a separate visit, completed three practice runs of a closed-circuit standardized course that included 8 driving maneuvers, followed by an on-road driving in the community fir 30 minutes.
  Interventions: Other: driving evaluation and practice
- drivers with normal cognition (Active Comparator): The participants firstly completed a questionnaire of driving history and perceived driving competence, followed with a clinical physical and cognitive-perceptual assessment battery conducted by an occupational therapist to note any potential deficits that might affect driving performance. The participants, on a separate visit, completed three practice runs of a closed-circuit standardized course that included 8 driving maneuvers, followed by an on-road driving in the community fir 30 minutes.
  Interventions: Other: driving evaluation and practice

INTERVENTIONS:
Other: driving evaluation and practice — The participants completed the actual driving with a licensed driving instructor on the passenger side in the car and with a dual-control, automatic-transmission car.
  Each participant completed three runs of the same route. The first twos were practices to familiarize themselves with the course. The driving instructor graded them on the third run. Each trial took about 10 minutes. The participants were scored according to governmental driver test guidelines. Scoring on individual driving maneuver is weighted. Depending on the type of error, 8, 16 or 32 points were deducted from 100, for example, 32 points for getting too close to pedestrian lane, running a red light or railroad crossing, and 8 points for stopping in S-curve forward and backward. 70 or above is considered as a pass. The occupational therapists in the backseat recorded driving behaviors, including whether the driver checked rear and side mirrors, excessive sweating, distractibility, number of adjustments, etc.

SUMMARY:
Driving is an important activity for older adults because it frequently relates to personal independence and wellbeing. This study compared the driving behaviors of older drivers with normal cognition and with MCI in unfamiliar driving situations and difficult maneuvers, and explored the practice effect on driving performance of drivers with MCI.

This study used an observational, cross-section research design.

DETAILED DESCRIPTION:
Driving is an important activity for older adults because it is frequently related to personal independence, mobility, social interaction, wellbeing, and confidence. Dementia can impair older adults' driving. The current consensus is that people with moderate or severe dementia are too cognitively impaired to drive safely. Persons with Mild Cognitive Impairment (MCI), often considered a transitional state to dementia, and those with mild dementia can still potentially drive, although some require further evaluation to determine the driver's fitness to drive. Extensive research has been devoted to the development of fitness-to-drive assessments. However, very limited attention has been paid to whether the driving skills of drivers with MCI can improve and thus potentially prolong the driver's safe-driving years.

MCI is a common neurodegenerative disease in older adults, with a prevalence of 16-20%. It is estimated that 20-40% of the MCI population will progress to dementia. Despite the potential driving concerns, it should be noted that over 50% of people with MCI are considered safe drivers. Because un-warranted driving cessation may lead to depression, functional decline, and even increases in the family's care burden, researchers have guarded against the premature revocation of driving rights.

Recent studies exploring the driving behaviors of drivers with MCI have shown inconsistent results. For example, increasing difficulties and unsafe behaviors in driving can be considered early warning signs of possible cognitive impairment. There may be a connection between specific cognitive skills (such as flexibility of visual attention and executive functioning) and poorer driving performance on specific tasks, such as car-following and road-tracking. Drivers with MCI may encounter difficulties at intersections with stop signs or critical light changes, and with headway, driving speed, reaction time, and lateral control. However, the above studies were usually conducted with driving simulators.

Only a few studies have investigated the on-road driving performance of drivers with MCI. Wadley, et al. compared drivers with MCI to drivers with normal cognition on a standardized route with various driving maneuvers frequently encountered in daily life. The results showed "less than optimal" performance, such as statistically significant poor performances in overall driving skills, especially in lane control and left turns. Driving can become increasingly difficult, for the cognitive capacities of older drivers with MCI are likely to deteriorate over time.

Recent evidence has suggested that cognitive training can slow or even reverse the cognitive impairments associated with MCI. Cognition intervention have shown positive improvements in the immediate and delayed memory functions of persons with MCI after intervention. However, advances in cognitive training for persons with MCI have yet to be applied to driver rehabilitation.

Driving rehabilitation includes both screening for unsafe drivers and the provision of individually-tailored interventions for clients with disabilities or those with a recent health event. Older drivers with cognitive impairments, such as dementia, are frequently the focus of driver screening. The current literature on driving training or retraining, however, has focused on other client populations, such as stroke, traumatic head injuries, and spinal cord injuries, and excluded those with cognitive impairments or not included screening for cognitive impairments. Even though systematic reviews by Korner-Bitensky et al. (2009) and Unsworth et al. (2014) support that driver rehabilitation improves the on-road driving performance of older drivers, older drivers with MCI are rarely considered targets for driver re-training. This finding is surprising because the driving skills of drivers with MCI can be compromised. Drivers with MCI can potentially benefit most from driving re-education, yet few studies have discussed issues related to driving training of older drivers with MCI.

In short, it is imperative to maintain the independence of persons with cognitive impairments for as long as possible. Without intervention, the driving competence of persons with MCI is likely to deteriorate as the disease and age progress. This study is to explore this possibility by examining how drivers with MCI perform as compared to drivers with normal cognition when negotiating a new route and whether learning effects would manifest if the drivers were given opportunities to practice.

ELIGIBILITY:
Inclusion criteria

* age of at least 50 years
* possession of a valid driving license and driving experience for at least 15 years
* regular driving habit, defined as at least once a week, and
* no reported significant driving issues

Exclusion Criteria

* reported health conditions that could potentially compromise driving competence, such as stroke, Parkinson's disease or other neuromuscular diseases
* visual impairments without correction, or
* physical impairments found in physical function assessments

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
driving evaluation | The participant was scored immediately after practices.
  The driving evaluation follows the same format of the governmental on-road driving tests in Taiwan. The test included 8 driving maneuvers on a standardized driving course: pre-drive checks and actions before starting to drive, crosswalk crossing, railway crossing, parking in reverse, parallel parking at roadside, driving forward and backward on a curving road (S-bend), ascending and descending slope, driving around the test circuit. https://tpcmv.thb.gov.tw/english/ServicesEng/LicenseEng/LicenseTest/t03.htm The participants were scored according to governmental driving licensure exam guidelines. Scoring on individual driving maneuver is weighted. Depending on the type of error, 8, 16 or 32 points were deducted from 100, for example, 32 points for getting too close to pedestrian lane. The minimal score is 0 and the maximal score is 100. Higher scores means better performance.
control of steering wheel | during the practices
  An Android smart phone (LG Nexus 5) was used to record on-road driving behaviors. The phone was equipped with a global positioning system (GPS) mobile application, J device. J device compiled the accelerator, gyroscope, and GPS data at a frequency of 50 Hz. The J device gyroscope data showed changes in driving direction, indicating whether the driver's control of the steering wheel was steady. Lower numbers in gyroscope data meant that the steering wheel was moved little, thus indicating few changes in direction or steadier hands on the steering wheel
control of speed | during the practices
  An Android smart phone (LG Nexus 5) was used to record on-road driving behaviors. The phone was equipped with a global positioning system (GPS) mobile application, J device (Tsao et al., 2015). J device compiled the accelerator, gyroscope, and GPS data at a frequency of 50 Hz. The J device accelerator data represented changes in the speed of the car, indicating the degree of control the driver had over the accelerator and brake; i.e., whether the driver maintained a steady speed or caused frequent changes in speed. A lower number of accelerations meant that the driver had smaller acceleration changes in a set period of time, indicating a more constant speed and thus better accelerator and brake control. A higher number of accelerations meant that the driver had larger acceleration changes in a set period of time, indicating greater variation in speed and less control of the accelerator and brake.

CONTACTS AND LOCATIONS:
Overall Officials: Ling-Hui Chang, Ph.D, Principal Investigator — Department of Occupational Therapy, NCKU

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheng YH, Pai MC, Shih BH, Jan SS, Lin CY, Chang LH. Driving practice effects for older drivers with mild cognitive impairment: A preliminary study. Scand J Occup Ther. 2023 May;30(4):550-558. doi: 10.1080/11038128.2023.2184420. Epub 2023 Mar 11. PMID 36905632